CLINICAL TRIAL: NCT04440241
Title: Regenerative Surgical Treatment of Peri-implant Defects. Submerged Versus Not Submerged
Brief Title: Regenerative Surgical Treatment of Peri-implant Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Osteology Foundation (Other)
Responsible Party: Principal Investigator, Juan Blanco Carrión, Principal investigator - Juan Blanco Carrión, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REGT_CT_19
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Implant Site Pocket Infection

STUDY DESIGN:
Intervention Model Description: Test group: submerged healing Control group: non-submerged healing treatment of peri-implantitis using guided bone regeneration with a bone substitute and a resorbable membrane.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): submerged healing treatment of peri-implantitis using guided bone regeneration with a bone substitute and a resorbable membrane.
  Interventions: Procedure: regenerative treatment periimplantitis
- Control group (Experimental): non submerged healing treatment of peri-implantitis using guided bone regeneration with a bone substitute and a resorbable membrane.
  Interventions: Procedure: regenerative treatment periimplantitis

INTERVENTIONS:
Procedure: regenerative treatment periimplantitis — Full thickness buccal and lingual flaps will be performed. After debridement of the defect using hand and ultrasonic instruments and implant surface decontamination using titanium brushes (TiBrush®) and saline Regenerative treatment will be performed only in the intrabony component of type 1 peri-implant defects. Guided bone regeneration using a bone substitute (Bio-oss®) and a resorbable membrane (bio-gide®) will be performed in the intrabony and dehiscenses areas of the defect.
  The surgeon will be blinded to the assignment of treatment until it is time to close the flaps.

SUMMARY:
Does submerged healing of implants improve clinical and radiologic outcomes for the treatment of peri-implantitis? A number of recent systematic reviews have shown that the prevalence of periimplantitisin the population is high.

Nevertheless, there appears to be no consensus on treatment standards for the management of peri-implant diseases. Also, the significant variation in the empirical use of the available therapeutic modalities seems to result in moderately effective treatment outcomes. Animal and human case series-studies have shown improved outcomes when using a submerged healing approach. However, there seems to be no randomized controlled clinical studies comparing submerged/non-submerged healing efficacy for the treatment of peri-implantitis. Since current modalities for the treatment of peri-implantitis seem to result inmoderately effective outcomes, there is an urgency to investigate treatment strategies that will result in improved patient's benefits in terms of health.

DETAILED DESCRIPTION:
The present study will be double-blinded randomized controlled clinical trial. Patients requiring surgical treatment of peri-implantitis after non-surgical therapy will beassigned to either:

Test group: submerged healing or Control group: non-submerged healing treatment of peri-implantitis using guided bone regeneration with a bone substitute and a resorbable membrane.

The primary aim of this study is to evaluate whether submerged healing of implants willsignificantly improve the changes in marginal bone levels measured on X-rays 12months post-treatment compared to a non-submerged healing approach for the treatment of peri-implantitis.

Secondary aims include changes in clinical attachment levels, changes in probing pocket depth, recession, keratinized tissue, occurrence of bleeding on probing, suppuration on probing (PUS), marginal gingival recession (REC), full mouth plaque score (FMPS), full mouth bleeding score (FMBS), type of peri-implant bone defect, frequency and type of complications and implant loss.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Systemically healthy patients.
* Presence of at least 1 implant diagnosed with peri-implantitis (peri-implant probing pocket depth ≥6 mm in at least 1 aspect of the implant with bleeding and/or suppuration on probing and radiographically documented marginal bone loss ≥3mm) according to Renvert et al. (2018), after non-surgical therapy of periimplantitis, and a 4mm deep intrabony component.
* Absence of mobility of the implants.
* Individual implant-supported crown or partial fixed implant supported restoration (removable prosthesis will be excluded).
* Patient's smoking ≤ 10 cigarettes/day.

Exclusion Criteria:

* Non-removable prostheses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes marginal bone level | baseline, 6 and 12 months
  measured on periapical X-rays, from the shoulder of the implant to the bottom of the bone defect next to the implant at the mesial and distal surfaces. Mean marginal bone levels between mesial and distal measurements will be calculated.

SECONDARY OUTCOMES:
Changes Probing pocket depth | baseline, 6 and 12 months
  distance from the margin gingival to the bottom of the peri-implant pouch. All clinical variables will be recorded with a Hu-friedy CP15 UNC millimeter probe in six points on each implant.
Changes Clinical attachment level | baseline, 6 and 12 months
  Distance from the implant shoulder or prosthetic abutment to the bottom of the peri-implant pocket.
Change Reccesion | baseline, 6 and 12 months
  distance from the margin of the peri-implant mucosa to the implant / abutment interface.
Change Keratinized mucosa | baseline, 6 and 12 months
  distance from the gingival margin up to the mucogingival line.
Change blending on probing | baseline, 6 and 12 months
  Registry of presence of bleeding by binary scale (1 bleed present / 0 bleed absent)
Change supuration | baseline, 6 and 12 months
  Pus presence register by scale binary (1 present / 0 absent)
Change plaque score | baseline, 6 and 12 months
  Registration of presence of plaque by binary scale on each surface (1 present / 0 absent), calculating the percentage of total surfaces in which plaque is detected by using a periodontal probe
configuration of the bone defect | baseline
  Based on the classification of Schwarz et al. (2007)

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Mareque, Study Director — University of Santiago de Compostela
Locations (1):
- Master Periodoncia. Facultad odontología, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schwarz F, Herten M, Sager M, Bieling K, Sculean A, Becker J. Comparison of naturally occurring and ligature-induced peri-implantitis bone defects in humans and dogs. Clin Oral Implants Res. 2007 Apr;18(2):161-70. doi: 10.1111/j.1600-0501.2006.01320.x. PMID 17348880
- [Result] Schwarz F, Sahm N, Schwarz K, Becker J. Impact of defect configuration on the clinical outcome following surgical regenerative therapy of peri-implantitis. J Clin Periodontol. 2010 May;37(5):449-55. doi: 10.1111/j.1600-051X.2010.01540.x. Epub 2010 Mar 24. PMID 20374416
- [Result] Roccuzzo M, Bonino F, Bonino L, Dalmasso P. Surgical therapy of peri-implantitis lesions by means of a bovine-derived xenograft: comparative results of a prospective study on two different implant surfaces. J Clin Periodontol. 2011 Aug;38(8):738-45. doi: 10.1111/j.1600-051X.2011.01742.x. Epub 2011 Jun 2. PMID 21635278